CLINICAL TRIAL: NCT01290393
Title: Post-marketing Safety Study to Assess the Risk of Spontaneous Abortion Following Administration of CERVARIX in the United States and Canada
Brief Title: Post-marketing Study to Assess the Safety of CERVARIX When Used in the United States and in Canada
Status: Terminated | Type: Observational
Why Stopped: Low accrual of subjects primarily attributable to the low uptake of Cervarix in the US and Canada in women aged 15 to 25 years of age.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The Organization of Teratology Information Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: 114176
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Infections, Papillomavirus
Keywords: vaccine; Spontaneous abortions; Human papillomavirus; HPV; Cervarix; pregnancy
MeSH Terms: conditions — Papillomavirus Infections; Abortion, Spontaneous | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Exposed vaccinated cohort: Women with last menstrual period between 30 days before and 90 days after any CERVARIX dose. The target sample size of the Exposed vaccinated cohort is 150 subjects.
  Interventions: Other: Data collection
- Non-exposed vaccinated cohort: Women with last menstrual period between 120 days and 18 months after the last CERVARIX or GARDASIL dose. The target sample size of the Non-exposed vaccinated cohort is 300 subjects.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection from hard copy interview forms routinely used by the Organization of Teratology Information Specialists (OTIS).

SUMMARY:
This study will assess the risk of spontaneous abortion during weeks 1-19 of gestation, and other pregnancy outcomes, in an Exposed vaccinated cohort, i.e. women with last menstrual period between 30 days before and 90 days after any dose of CERVARIX, when compared to a Non-exposed vaccinated cohort, i.e. women with last menstrual period between 120 days and 18 months after the last CERVARIX or GARDASIL dose.

DETAILED DESCRIPTION:
The present study will be conducted by the OTIS (Organization of Teratology Information Specialists) network. OTIS is a non-profit organization specialised to assess exposures during pregnancy and dedicated to providing accurate evidence-based, clinical information to patients and health care professionals about exposures during pregnancy and lactation. OTIS is based on voluntary phone calls. Women call when they have questions and concerns about risks potentially associated with any kind of exposure during pregnancy or breastfeeding, including medications, chemicals, pesticides, diseases, infections, and vaccinations.

ELIGIBILITY:
Inclusion Criteria:

For Exposed vaccinated cohort:

* Written informed consent, and assent in case of minors, obtained from the subject/from the parent(s)/legally acceptable representative(s) of the subject.
* Aged between, and including, 15 and 25 years of age.
* Residing within the US or Canada.
* Subjects who received at least one dose of CERVARIX.
* Gestational age at inclusion should be 19 completed weeks (i.e. 133 days of gestation) or less.
* Last menstrual period between 30 days before and 90 days after any dose of CERVARIX with a maximum of 20% of subjects with last menstrual period between 46 and 90 days after any dose of CERVARIX.
* Subjects who the Investigator believes can and will comply with the requirements of the protocol (e.g. available for phone interviews). Or subjects who the Investigator believes that parent(s)/legally acceptable representative(s) can and will comply with the requirements of the protocol.

For Non-exposed vaccinated cohort:

* Written informed consent, and assent in case of minors, obtained from the subject/from the parent(s)/legally acceptable representative(s) of the subject.
* Aged between, and including, 15 and 25 years of age.
* Residing within the US or Canada.
* Subjects who received at least one dose of CERVARIX or at least one dose of GARDASIL.
* Gestational age at inclusion should be 19 completed weeks (i.e. 133 days of gestation) or less.
* Last menstrual period between 120 days and 18 months after the last dose of CERVARIX/ GARDASIL.
* Subjects who the Investigator believes can and will comply with the requirements of the protocol (e.g. available for phone interviews). Or subjects who the Investigator believes that parent(s)/legally acceptable representative(s) can and will comply with the requirements of the protocol.

Exclusion Criteria:

For Exposed vaccinated cohort:

* Last menstrual period between 30 days before and 90 days after any GARDASIL dose.
* Ongoing pregnancy with foetus known to be non-viable.
* Ongoing pregnancy with pre-enrolment knowledge by prenatal diagnosis of a major structural defect.
* Use of any investigational or non-registered product (drug or vaccine) during the study period.

For Non-exposed vaccinated cohort:

* Ongoing pregnancy with foetus known to be non-viable.
* Ongoing pregnancy with pre-enrolment knowledge by prenatal diagnosis of a major structural defect.
* Use of any investigational or non-registered product (drug or vaccine) during the study period.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women aged 15 to 25 years and residing in the United States or in Canada
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2012-12-20 (Actual); Study Completion 2012-12-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of spontaneous abortion during weeks 1-19 of gestation | This outcome measure will be recorded between zero and six weeks after end of pregnancy

SECONDARY OUTCOMES:
Occurrence of other adverse pregnancy outcomes | This outcome measure will be recorded between zero and six weeks after end of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, San Diego, California, United States